CLINICAL TRIAL: NCT04720248
Title: Valoración Del Dolor Postoperatorio en Pacientes Sometidos a craneotomía Programada
Brief Title: Postoperative Pain in Scheduled Craniotomy
Status: Completed | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Ángel Becerra, Principal Investigator, Dr. Negrin University Hospital
Other Study IDs: Craneo-Negrín
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Pain, Postoperative; Craniotomy; Adverse Effect; Anxiety
Keywords: postoperative pain; neurosurgery; craniotomy; anxiety
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders | interventions — Dipyrone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Metamizol postoperatively: Patients submitted to scheduled craniotomy receiving metamizol as analgesic medication postoperatively
  Interventions: Drug: Metamizole
- Paracetamol or other analgesics postoperatively: Patients submitted to scheduled craniotomy receiving paracetamol or other drugs as analgesic medication postoperatively

INTERVENTIONS:
Drug: Metamizole — Patients will receive metamizole intraoperatively and throughout 48h postoperatively.
  Groups: Metamizol postoperatively

SUMMARY:
Postoperative pain after craniotomy is frequent, with moderate-severe intensity. The fear to the side effects of opioids (nausea and vomiting and sedation), and NSAIDs (bleeding) makes it difficult to obtain adequate analgesic control in these patients. Preoperative anxiety may be associated with a poorer postoperative analgesic control, hindering the adequate postoperative evolution and increasing hospital stay and adverse effects. In this observational study, the investigators aimed to assess the postoperative analgesic management in patients undergoing scheduled craniotomy following routine clinical practice and to relate preoperative anxiety with the postoperative analgesic evaluation in this population.

DETAILED DESCRIPTION:
Postoperative pain after craniotomy is frequent, with moderate-severe intensity. The fear to the side effects of opioids (nausea and vomiting and sedation), and NSAIDs (bleeding) makes it difficult to obtain adequate analgesic control in these patients. On the other hand, preoperative anxiety may be associated with a poorer postoperative analgesic control and hinder the adequate postoperative evolution. The main outcome is to assess the postoperative analgesic management in patients undergoing to craniotomy. Secondary objectives are to evaluate the appearance of postoperative side effects related to the analgesics and to assess the relationship between preoperative anxiety and postoperative pain

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old undergoing scheduled form for supratentorial craniotomy.
* Signed informed consent.

Exclusion Criteria:

* Mini Mental State Examination with a score less than or equal to 24 points.
* Patients suffering from disabilities.
* Patients who can not collaborate in the postoperative clinical assessment.
* Patients who can not be assessed during the postoperative period by the Acute Pain Unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old undergoing scheduled form for supratentorial craniotomy during the 8 months following the beginning of study at the center who can give informed consent and can be postoperatively evaluated by the acute pain unit.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 48 hours postoperatively
  Using the Visual Analgesic Scale (from 0 to 10, with 0 being the state corresponding to "no pain" and 10 being the "maximum pain imaginable ") and postoperative analgesic satisfaction assessed by the patient (stratified in Bad, Fair, Good or Excellent).

SECONDARY OUTCOMES:
Side effects secondary to metamizol | 48 hours postoperatively
  Rate of appearance of postoperative side effects.
To assess the correlation between preoperative anxiety and postoperative pain. | From the day before surgery to the second day postoperatively
  Relate the score obtained in the State Anxiety Inventory Trait (STAI) (from 0 to 60) with the intensity of postoperative pain (from 0 to 10).

CONTACTS AND LOCATIONS:
Overall Officials: Aurelio Rodríguez Pérez, PhD, Study Director — Hospital Universitario de Gran Canaria Doctor Negrín; Ángel Becerra, MD, Principal Investigator — Hospital Universitario de Gran Canaria Doctor Negrín
Locations (1):
- Ángel Becerra, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be decided to be available to other researchers once the study ends.